CLINICAL TRIAL: NCT05444361
Title: Eliminating Post-Mastectomy Pain and Opioids With Percutaneous Cryoneurolysis: A Single-Administration, Non-Opioid, Non-Addictive, Multiple-Month Analgesic
Brief Title: Ultrasound-Guided Percutaneous Cryoneurolysis to Treat Postoperative Pain After Mastectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Department of Defense Congressionally Directed Medical Research Program (Unknown)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRYO for Mastectomy (DoD)
Record Dates: First submitted 2022-06-24; First posted 2022-07-05 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Mastectomy; Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: Pragmatic, multicenter, randomized, triple-masked, sham-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators, participants, and clinical staff will be masked to treatment group assignment, with the only exception being the unmasked individual who performs the procedure (and will not have subsequent contact with the participant).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoneurolysis (Active Comparator): Cryoneurolysis of the 2nd-6th thoracic intercostal nerves will be treated on the ipsilateral surgical side (bilaterally for bilateral surgical procedures): for each nerve the cryoneurolysis device will be triggered using 1 cycle of 5.5-minute [all but 4 participants: 064-067] or 3 minutes [only 4 participants 064-067; change based on new laboratory data, then changed back based on inadequate freeze] argon activation (2000 psi and 100% power) followed by a 30-second helium defrost. For active probes, the gas will be deployed to the tip where a drop in temperature to approximately -70°C will result in cryoneurolysis.
  Interventions: Device: Cryoneurolysis
- Sham Procedure (Sham Comparator): Sham cryoneurolysis of the 2nd-6th thoracic intercostal nerves will be applied on the ipsilateral surgical side (bilaterally for bilateral surgical procedures): for each nerve the cryoneurolysis device will be triggered using 2 cycles of 2-minute gas activation separated by 1-minute defrost periods (Epimed) or 1 cycle of 5.5 minutes [all but 4 participants: 064-067] or 3 minutes [only 4 participants 064-067; change based on new laboratory data, then changed back based on inadequate freeze] of argon and 30 seconds of helium (Varian). However, for sham probes, the gas is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Cryoneurolysis — Cryoneurolysis of the 2nd-6th thoracic intercostal nerves will be treated on the ipsilateral surgical side (bilaterally for bilateral surgical procedures): for each nerve the cryoneurolysis device will be triggered using 2 cycles of 2-minute gas activation separated by 1-minute defrost periods (Epimed) or 1 cycle of 5.5 minutes [all but 4 participants: 064-067] or 3 minutes [only 4 participants 064-067; change based on new laboratory data, then changed back based on inadequate freeze] of argon and 30 seconds of helium (Varian). For active probes, the gas will be deployed to the tip where a drop in temperature to approximately -70°C will result in cryoneurolysis.
  Other Names: Cryoablation
  Arms: Cryoneurolysis
Device: Sham Comparator — Sham cryoneurolysis of the 2nd-6th thoracic intercostal nerves will be applied on the ipsilateral surgical side (bilaterally for bilateral surgical procedures): for each nerve the cryoneurolysis device will be triggered using 2 cycles of 2-minute gas activation separated by 1-minute defrost periods (Epimed) or 1 cycle of 5.5 minutes [all but 4 participants: 064-067] or 3 minutes [only 4 participants 064-067; change based on new laboratory data, then changed back based on inadequate freeze] of argon and 30 seconds of helium (Varian). However, for sham probes, the gas is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Other Names: Sham procedure
  Arms: Sham Procedure

SUMMARY:
Breast cancer is the most common type of cancer in women. Removal of the breast, called "mastectomy", is performed either when there is cancer-or an increased risk of cancer-in the breast. This can result in a lot of pain during the months after surgery. Opioids-"narcotics"-are the most common pain control method provided to patients; but they frequently do not relieve enough pain, have undesirable side effects like vomiting and constipation, and are sometimes misused which can lead to addiction. Mastectomy also frequently results in long-term pain which can interfere with physical and emotional functioning; and the more pain patients have immediately after surgery, the greater the risk of developing long-term pain. Numbing the nerves with local anesthetic can decrease the amount of short- and long-term pain experienced by patients, but even the longest types of these nerve blocks last for hours or days, and not the 1-2 months of pain typically following mastectomy. So, there is reason to believe that if the nerve blocks could be extended so that they last longer than the pain from surgery, short- and long-term pain might be avoided completely without the need for opioids. A prolonged nerve block may be provided by freezing the nerve using a technique called "cryoneurolysis". With cryoneurolysis and ultrasound machines, a small needle-like "probe" may be placed through anesthetized skin and guided to the target nerve to allow freezing. The procedure takes about 5 minutes for each nerve, involves little discomfort, has no side effects, and cannot be misused or become addictive. After 2-3 months, the nerve returns to normal functioning. The investigators have completed a small study suggesting that a single cryoneurolysis treatment may provide potent pain relief after mastectomy. The ultimate objectives of the proposed research study are to determine if temporarily freezing the nerves that go to the breast will decrease short-term pain, opioid use, physical and emotional dysfunction, and long-term pain following mastectomy when added to current and customary postoperative analgesics.

The current project is a pragmatic, multicenter, randomized, triple-masked (investigators, participants, statisticians), sham/placebo-controlled, parallel-arm, human-subjects, post-market clinical trial to determine if cryoneurolysis is an effective non-opioid treatment for pain following mastectomy.

DETAILED DESCRIPTION:
All participants will continue to receive standard and customary postoperative analgesics of their local treatment center, so there is no risk of participants receiving a lower degree of analgesia than if they otherwise did not enroll in the study. The cryoneurolysis procedure will be done in addition to standard local institutional standard analgesic treatments.

The investigators propose a pragmatic, multicenter, randomized, triple-masked (investigators, participants, statisticians), sham/placebo-controlled, parallel-arm, human-subjects clinical trial to determine if cryoneurolysis is an effective non-opioid treatment for pain following mastectomy. Participants will be individuals undergoing unilateral or bilateral mastectomy, recruited at 6 centers:

* Walter Reed National Military Medical Center, Bethesda, Maryland
* U.C. San Diego, San Diego, California
* University of Florida, Gainesville, Florida
* Cedars-Sinai, Los Angeles, California
* Cleveland Clinic, Cleveland, Ohio

For women of childbearing age with the possibility of pregnancy, a sample of urine will be collected before any study interventions to confirm a non-pregnant state. Participants will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied (blood pressure cuff, pulse oximeter, 5-lead ECG), and oxygen administered via a facemask. Midazolam and fentanyl (IV) will be titrated for patient comfort as needed throughout the procedure, while ensuring that patients remain responsive to verbal cues.

Peripheral nerve block. Not all enrolling centers provide peripheral blocks as part of their standard-of-care. Due to the pragmatic design of this trial, study participation will not alter an institution's current practice. If the local practice includes a postoperative continuous peripheral nerve block, a perineural catheter will be inserted 2-5 cm beyond the needle tip, the needle withdrawn over the catheter, the catheter affixed with an occlusive sterile dressing.

Participants will be allocated to one of two treatments:

1. cryoneurolysis
2. sham cryoneurolysis (placebo control)

Randomization will be stratified by enrolling institution, surgical site (unilateral vs. bilateral), and axillary involvement (none/biopsy vs. dissection) in a 1:1 ratio, and in randomly chosen block sizes. Randomization lists will be created using Statistical Analysis Software computer-generated tables by the informatics division of the Department of Outcomes Research (Cleveland Clinic, Cleveland, OH). Treatment group assignment will be conveyed to the enrolling sites via the same secure web-based system (REDCap) used to collect and collate all post-intervention endpoints.

There are multiple types of cryoneurolysis machines cleared by the US FDA, all of which work on the same principle of a gas being passed through a small annulus, resulting in a dramatic pressure drop and accompanying temperature drop due to the Joule-Thomson effect. This study will utilize two different consoles [second option added May 8, 2023]: the Epimed International (Farmers Branch, TX) and Varian Medical Systems (Palo Alto, CA) machines. Which machine is used is determined simply by the machine that each enrolling center has at its disposal.

Varian: This machine uses argon for the freeze cycle and helium to help decrease the thaw period duration. Sham probes are not available for this type of machine, and therefore an active probe will be used for all participants. For participants randomized to active treatment, the probe will be connected to the machine as usual, the argon (and helium) passed through the probe and then back into the machine, and finally vented out from the console. For participants randomized to sham treatment, the probe will be connected to an inactive connector on the back of the machine. For these participants the gas will simply be ejected directly from the console without ever having passed through the probe. The investigator administering the study intervention will access the treatment group assignment using the secure web-based system and attach the probe (active) or leave the tubing end close to the machine (sham). Therefore, all investigators, participants, and clinical staff will be masked to treatment group assignment, with the only exception being the unmasked individual who performs the procedure (and will not have subsequent contact with the participant).

Epimed: This machine uses nitrous oxide for the freeze cycle with a passive thaw (no gas flow). Cryoneurolysis probes are available that either (1) pass nitrous oxide to the distal end inducing freezing temperatures; or (2) vent the nitrous oxide at the proximal end of the probe so that no gas reaches the distal end, resulting in no temperature change. The latter is a sham procedure since without the temperature change, no ice ball forms and therefore the target nerve is not affected. Importantly, these probes are indistinguishable in appearance and will be differentiated only by an identifying stamp on the underside of the connector which is not visible during use.

The investigator administering the study intervention will access the treatment group assignment using the secure web-based system and attach the appropriate probe to the cryoneurolysis device. Therefore, all investigators, participants, and clinical staff will be masked to treatment group assignment, with the only exception being the unmasked individual who performs the procedure (and will not have subsequent contact with the participant). For both types of machines, it is impossible to mask the individual performing the cryoneurolysis procedure because the ice ball forming at the distal end of the probe-with active treatment-is clearly visible by ultrasound; and the lack of an ice ball for placebo participants is equally clear. It is essential to continuously visualize the probe and target nerve throughout the freeze/thaw cycle(s) to ensure the entire nerve diameter is adequately treated and remains relatively motionless. This cannot be achieved if the ultrasound is turned off during gas administration in an attempt to mask the provider.

Study intervention. The 2nd-6th thoracic intercostal nerves will be treated on the ipsilateral surgical side (bilaterally for bilateral surgical procedures). Using a curved-array transducer, the intercostal nerve will be visualized using ultrasound just inferior to each treated rib immediately distal to the costotransverse joint. For participants without a paravertebral block, a skin wheal of lidocaine 1% will be raised immediately inferior to the transducer to anesthetize the skin. An IV-like hollow-bore introducer may be inserted through the skin and guided to the target nerve--this is based on operator personal preference. For participants without anesthetized intercostal nerves from a peripheral nerve block, lidocaine 1.5-2.0% 2 mL may be injected through the introducer prior to the cryoneurolysis probe introduction to provide anesthesia during the cryoneurolysis cycles, although this is not universally applied (they cryoneurolysis treatment itself induces anesthesia).

A portable cryoneurolysis device (Varian CryoCare or Epimed PainBlocker) will be used. The probe will be inserted adjacent to the intercostal nerve.

Varian: The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute [all but 4 participants: 064-067] or 3 minutes [only 4 participants 064-067; change based on new laboratory data, then changed back based on inadequate freeze] argon activation (2000 psi and 100% power) followed by a 30-second helium defrost.

Epimed: The cryoneurolysis device will be triggered using 2 cycles of 2-minute gas activation (active or sham) separated by a 1-minute defrost.

The introducer and probe will be withdrawn and this process repeated for each additional intercostal nerve to be treated. For bilateral mastectomies, the study intervention will be repeated on the contralateral side with the same probe.

Intraoperative course. Due to the pragmatic nature of this trial, the investigators aim to change each center's standard practice as little as possible and rather investigate the results of adding the intervention to current practice. The investigators will therefore record intraoperative factors such as type of general anesthetic, axillary dissection, opioid administration, and local anesthetic supplementation; however, the investigators will not require changes to current standard practice.

Postoperative course. Standard local supplemental analgesics will be used due to the pragmatic design of this trial. For analysis purposes, all opioids will be converted to oral oxycodone equivalents. Following a cryoneurolysis treatment, no action is required by patients regarding this intervention. For example, in contrast to epidural infusions, there is no infusion pump to manage or anesthetic fluid to replenish. At enrolling centers that provide a postoperative continuous peripheral nerve block, the ropivacaine or bupivacaine infusions will be administered per local protocol with the catheters removed on postoperative day 1 or 2 prior to hospital discharge.

Following study completion, the results will be mailed electronically or by the United States Postal Service to all enrolled participants in written form using non-technical (e.g., "layperson") language.

Outcome Measurements (End Points). The investigators have selected outcome measures that have established reliability and validity, with minimal inter-rater discordance, and are recommended for pain-related clinical trials by the World Health Organization and the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consensus statement (Table 1, below).5 End points will be evaluated at baseline (prior to surgery on postoperative day 0), as well as postoperative days 1, 2, 3, 4, 7, 21, 30, 45; and months 2, 3, 6, 9 and 12).

Statistical Plan and Data Analysis

Primary Specific Aim: To determine the effect of cryoneurolysis on postoperative opioid requirements and analgesia following mastectomy.

Hypothesis 1: Opioid consumption will be significantly decreased in the first two months following surgery with cryoneurolysis compared with usual and customary analgesia.

Hypothesis 2: Surgical pain will be significantly decreased within the first two months following surgery with cryoneurolysis compared with usual and customary analgesia (measured with a Numeric Rating Scale).

Primary end point: In order to claim that cryoneurolysis is superior to usual and customary analgesia, at least one of Hypotheses 1 and 2 above must be superior while the other at least noninferior.

Secondary Specific Aims: To determine the effect of cryoneurolysis on physical and emotional functioning and chronic pain following mastectomy.

Hypothesis 3: Physical and emotional functioning will be significantly improved within the first two months following surgery with cryoneurolysis as compared with usual and customary analgesia (measured with the Interference Domain of the Brief Pain Inventory).

Hypothesis 4: The incidence of chronic pain will be significantly decreased 6 and 12 months following surgery with cryoneurolysis as compared with usual and customary analgesia.

Hypothesis 5: The intensity of chronic pain will be significantly decreased 6 and 12 months following surgery with cryoneurolysis as compared with usual and customary analgesia (measured with a Numeric Rating Scale).

Balance on baseline covariates will be assessed using absolute standardized difference (ASD):50 i.e., difference in means or proportions divided by the standard deviation. ASD > 0.1 will be considered to indicate imbalance, and these variables will be adjusted for in the statistical analyses. Analyses will be carried out using modified intention-to-treat (i.e., patients who received any study treatment will be analyzed according to the group to which they were randomized). The overall type I error rate of the study will be controlled using a parallel gatekeeping procedure (see Study-wide Type I error rate control).

Primary Objective (Hypotheses 1 and 2). The investigators will estimate the treatment effect of cryoneurolysis on opioid consumption (Hypothesis 1) and average pain score (Hypothesis 2) using a joint hypothesis-testing framework. The investigators will conclude that cryoneurolysis is more effective compared to the standard of care if it is noninferior on both opioid consumption and pain score, and superior for at least one of the outcomes during the first 2 months after surgery. No adjustment for multiple testing is needed for noninferiority testing since the investigators require noninferiority on both pain score and opioid consumption outcomes.

Noninferiority Testing.

Hypothesis 1 (Opioid consumption). Cumulative opioid assumption is typically log-normally distributed. The investigators will therefore assess the treatment effect on the log-transformed cumulative opioid consumption at 2 months using a linear regression model. The investigators will test for NI of cryoneurolysis to standard of care using a 1-tailed test assuming alpha of 0.025 and NI delta of 1.2 for the ratio of geometric means (treatment/placebo). All opioids will be converted to oral oxycodone equivalents.

Hypothesis 2 (Average pain score). The investigators will test for noninferiority (NI) of cryoneurolysis to standard of care using 1-tailed tests and assuming a 1-tailed alpha of 0.025. The primary pain outcome will be the area under the curve (AUC) of patient "average" pain scores over the first 2 months (60 days; AUC-60). For this outcome the noninferiority (NI) delta will be a ratio of geometric means of 1.2 in the AUC-60. Since AUC-60 is expected to be skewed and to have some proportion of zero values, the investigators will estimate the treatment effect a 2-sample t-test on the log-transformed (AUC-60 + 1). Noninferiority will be concluded if the upper 95% confidence interval of the ratio of geometric means is below the NI delta.

Superiority Testing. If NI is found on both pain and opioid use, the investigators will test for superiority on each of cumulative opioid consumption and average pain AUC-60 using 1-tailed tests (using the primary analyses specified above) with overall 1-tailed alpha of 0.025. Since there are 2 tests for superiority the investigators will apply a Holm-Bonferroni correction and use a significance criterion of 0.025/2 for the smaller P-value and 0.025 for the larger. Similar tests will be conducted for the sensitivity analyses for pain score. Cryoneurolysis will be concluded more effective at pain management than standard care, and the joint null hypothesis rejected, if found superior on at least pain score or opioid consumption and at least noninferior on both.

Secondary pain outcomes in first 60 days. For each of average, current, least and worst pain score, as well as the pain with ipsilateral arm raise, the investigators will conduct all of the analyses describe above for average pain score, as well as 1) assessing the treatment-by-time interaction in a linear mixed effects model using all measurements over time, and 2) estimating and reporting the treatment effect at each time point while controlling type I error across time points within each outcome variable using the Holm-Bonferroni procedure.

Sensitivity analyses for average pain score methodology. In addition to analyzing the AUC, the investigators will assess the treatment effect on patient "average" pain scores over time using a linear mixed effects model assuming an autoregressive (AR[1]) correlation structure across scores for the same individual over time. Factors will be intervention, time (categorical) and baseline average pain score. The investigators will then test for noninferiority with a 1-tailed t-test in which the numerator is the estimated treatment effect minus the NI delta of 1 point and the denominator is the standard error of the estimated treatment effect. In another sensitivity analysis, the investigators will use a mixed effects proportional odds model with an autoregressive correlation structure to assess the treatment effect on pain score as an ordinal outcome.

Hypothesis 3 (Physical and emotional functioning). Physical and emotional functioning of patients will be assessed using: 1) the interference domain of the Brief Pain Inventory (BPI), and 2) the Patient Health Questionnaire (PHQ-2). For the BPI Interference subscale, the effect of the intervention will be assessed over the first 2 months as in Hypotheses 2 and 3 -- using patient AUC as primary analysis and a linear mixed model adjusting for baseline BPI-Interference domain score as secondary. The investigators will further analyze the outcome over the entire first 12 months in a linear mixed effects model and compare the treatment groups at each time point, controlling type I error as specified in the primary objective under "Secondary pain outcomes in first 60 days". The effect of the intervention on depression as assessed by the Patient Health Questionnaire (PHQ-2) at 3-12 months will be analyzed by Wilcoxon rank-sum tests at each time, with treatment effect estimated as median difference (95% CI).19,20 In addition, a proportional odds logistic regression analysis adjusting for clinical site will be conducted for each time point.

Hypotheses 4 and 5 (chronic pain). The effect of the intervention on the maximum/worst pain (ordinal scale) experienced by patients at each of 6 and 12 months will be assessed by separate Wilcoxon rank-sum tests at each time point, with treatment effect estimated as median difference (95% CI). In addition, a proportional odds logistic regression analysis adjusting for clinical site will be conducted for each time point. Second, the effect of the intervention on presence of any pain (binary - yes/no) at each of 6 and 12 months will be assessed using chi-square analyses and relative risk (95% CI), as well as Cochran-Mantel-Haenszel tests stratified by clinical site.

Study-wide Type I error control. The investigators will use a parallel gatekeeping procedure to control the study-wide type I error at 0.05. For this procedure the investigators therefore have prioritized (a priori) the study outcomes into 7 ordered sets (Table 5, following page). Analysis will proceed in that order, and testing will proceed through each "gate" to the next set if and only if at least one outcome in the current set reaches significance. The significance level for each set will be 0.05 times a cumulative penalty for non-significant results in previous sets (i.e., a "rejection gain factor" equal to the cumulative product of the proportion of significant tests across the preceding sets). Within a set, a multiple comparison procedure (Holm-Bonferroni correction) will be used as needed to control the type I error at the appropriate level. Although the first set represents the 1-tailed joint hypothesis tests for noninferiority and superiority at alpha=0.025, without modifying the joint hypothesis test the investigators will use the corresponding 2-tailed alpha level of 0.05 for the gatekeeping, as all other sets involve 2-tailed tests. Some of the outcomes listed in the gatekeeping table are overall assessments over repeated measures. As detailed in statistical methods, treatment effects may also be assessed at individual time points. Such assessments will proceed according to the gatekeeping framework such that 1) type I error will be controlled across repeated measurements, and 2) inference will not be made on outcome variables that are excluded from formal testing/inference due to the gatekeeping results.

Parallel gatekeeping procedure [revised December 12, 2022, after 7 participants were enrolled because the study is a pragmatic trial and not all enrolling centers include peripheral nerve blocks and/or perineurial local anesthetic infusions as part of their standard care; and therefore anticipated opioid consumption and pain scores will be higher across all groups relative to the single-center pilot study]

Sets: Time frame... Required to pass to next set

1. H1/H2 - Joint hypothesis - opioids and pain Requires: NI both, superiority on at least one, 2 months, Reject joint H0 (1 joint test)
2. H3 - BPI interference subscale, 2 months, Significance on this outcome
3. H4/H5 - Chronic pain: (1) incidence and (2) worst pain, 6 months, Significance on either outcome H4/H5
4. H4/H5 - Chronic pain: (1) incidence and (2) worst pain, 12 months, Significance on either outcome H4/H5
5. H2 - Percentage of each group that required <=3 opioid tablets from recovery room discharge through 2 mos
6. H1 - Percentage of each group that experienced no more than moderate (NRS < 7) pain at all time points 2 months, Significance on either outcome 5 or 6
7. H3 - Depression screen PHQ-2 6 & 12 months Significance on either outcome

Interim Analyses. The investigators will use a group sequential design with a non-binding futility boundary and conduct an interim analysis at 50% of the maximum planned enrollment to assess the efficacy/futility of the intervention. Specifically, the investigators will maintain the overall alpha level (monitoring efficacy) at 0.025 using gamma parameter of -4 and power at 90% (monitoring beta, type II error) using gamma parameter of -4. Under the alternative hypothesis, the cumulative probability of crossing an efficacy (and futility in parentheses) boundary at the 1st and 2nd analyses will be 0.33 (0.01), and 0.90 (0.10). Under the joint hypothesis testing framework, the investigators aim to have 90% power to detect NI on both outcomes and superiority on any one outcome.

Sample Size Justification and Power Analyses. Sample size calculations and power analyses for the full study were informed by estimates from the pilot trial. The investigators plan to have 90% power for rejecting the joint hypothesis test for the primary aim.

Opioids. In the pilot study (N=30), the median [quartiles] of cumulative opioid consumption over 60 days was 91 [15, 146] in the control group and 3 [0, 15] in the treatment group. The ratio of geometric means [95% CI] was 0.13 [0.03, 0.54] indicating an 87% estimated relative percent reduction in cumulative opioid consumption at 60 days. The investigators observed a coefficient of variation (CV) of 1.4. Noninferiority: Assuming a geometric mean ratio of 0.70, a NI delta of 1.2, alpha of 0.025 and CV of 1.4, the investigators would have 96.2% power to reject the null hypothesis. Superiority: A sample size of 108 patients in each group would yield 95.0% power to detect a geometric mean ratio of 0.57 (treatment/ placebo), assuming a CV of 1.4, a 1-tailed alpha of 0.0125, and after adjusting for interim analyses.

Pain. In the pilot study (N=30), the median [quartiles] of AUC-60 was 29 [16, 67] in the control group and 1 [0, 4] in the treatment group. The ratio of geometric means [95% CI] was 0.10 [0.04, 0.27] indicating a 90% estimated relative percent reduction in pain score at 60 days in treatment versus placebo. The investigators observed a coefficient of variation (CV) of 1.4. Noninferiority: Assuming a true ratio of geometric means in AUC-60 of 0.71, a NI delta of 1.2, a 1-tailed alpha of 0.025 and CV of 1.4, a sample size of 108 patients per group would yield 95.3% power to detect noninferiority of cryoanalgesia versus control after adjusting for interim analyses. Superiority: A sample size of 108 patients in each group would yield 95.0% power to detect a geometric mean ratio of 0.57 (treatment/placebo), assuming a CV of 1.4, a 1-tailed alpha of 0.0125, and after adjusting for interim analyses. With the same sample size, the investigators would have 92.4% power to detect a decrease of 1 point in the pain score assuming alpha = 0.0125, standard deviation of 2.5, intraclass correlation coefficient (ICC) of 0.55 and an average cluster size (measurements per participant) of 7.

Power for Joint Hypothesis test. The investigators will have 90% power to reject the joint null hypothesis, e.g., 95% power for superiority on pain score times 96% power for noninferiority on opioids = 91%, assuming independence between the two outcomes.

Loss to follow-up. Within our pilot study (n=30) there were no lost patients for the full 1-year follow-up period. However, this might be a unique subset of patients which may differ from a future cohort at the same or other enrolling centers. Based on previous multicenter clinical trials, the investigators estimate that at most 7% of participants in each group are expected to drop out of the study before reaching the 2-months primary outcome assessment. For those missing data the investigators will use intent-to-treat and multiple imputation (multiple imputation for chained equations (MICE)) using data on all observed baseline and outcome data.

Sample size re-estimation. At the first interim analysis (50% of maximum enrollment), the investigators will estimate variance and ICC of the pain scores, and CV for opioids, and re-estimate the required sample size. All analyses will either adjust for clinical site (e.g., in a regression model) or consider it as a stratification variable (e.g., in a Cochran-Mantel-Haenszel relative risk analysis). Statistical Analytic Software (Carey, North Carolina), R programming language (The R Project for Statistical Computing) and East 5.3 software (Cytel Inc.) will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of at least 18 years of age
2. Undergoing unilateral or bilateral total or modified radical mastectomy

Exclusion Criteria:

1. Anticoagulation or bleeding disorder: introduction of the percutaneous cryoneurolysis probe has a risk of hemorrhage similar to the percutaneous insertion of a similar gauge needle; but an anticoagulated state will increase the risk of hemorrhage (aspirin in doses for cardiothoracic/stroke prophylaxis [≤ 325 mg] are acceptable).
2. Infection at the site of probe introduction: percutaneous insertion of the probe through a cutaneous infection would bring an unacceptable risk of introducing the infection to deeper tissues.
3. Pulmonary disease requiring supplemental oxygen: one theoretical risk of cryoneurolysis is a unilateral pneumothorax (not reported) which could result in a compromised pulmonary state for patients who require supplemental oxygen at baseline.
4. Possessing any contraindication to decreased temperature such as cryoglobulinemia, cryofibrinogenemia, cold urticaria, paroxysmal cold hemoglobinuria, or Raynaud's disease: the decreased temperature accompanying cryoneurolysis could result in local tissue/vascular compromise for patients with any of these cold-triggered syndromes/diseases.
5. Neurologic deficit of the 2nd-6th ipsilateral intercostal nerves: cryoneurolysis is theoretically a potent analgesic, but it does not "heal" injured nerves. Therefore, pre-existing nerve deficits will confound the analgesia-related results.
6. Chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks, either by self-report or recorded previously in the medical record): individuals using opioids on a chronic basis will continue their baseline opioid requirements postoperatively. This will confound the analgesic results of the study.
7. Insulin-dependent diabetes: laboratory studies have demonstrated impaired nerve regeneration in diabetic animals, and diabetes in patients can lead to impaired regeneration of axons and recovery following investigational nerve injury65 as well as focal neuropathies such as ulnar neuropathy and carpal tunnel syndrome. Whether these findings are applicable to cryoneurolysis in patients with diabetes remains unknown, but we prefer to err on the side of caution for study participants.
8. Contralateral breast surgical procedure that does not include mastectomy.
9. Inability to remain in contact with the investigators during the study period (e.g., lack of telephone access).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-05-14 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption during first 2 postoperative months | Postoperative months 1 and 2, collected on days 1, 2, 3, 4, 7, 14, 21, 30, 45 and 60; at each collection time point, opioid use for the previous 24 hours will be recorded
  Cumulative opioid dose measured in oral oxycodone equivalents following recovery room discharge for 10 specific 24-hour time points over the first 2 months following surgery. With 10 time points (postoperative days 1, 2, 3, 4, 7, 14, 21, 30, 45 and 60), this will encompass 240 hours in total of the first 2 postoperative months. In order to claim that percutaneous cryoneurolysis is superior to usual and customary analgesia, at least one of Outcomes 1 and 2 must be superior while the other at least noninferior.
Average pain during first 2 postoperative months | Postoperative months 1 and 2, collected on days 1, 2, 3, 4, 7, 14, 21, 30, 45 and 60; at each collection time point, the "average" pain score for the previous 24 hours will be recorded
  The area under the curve for the "average" daily pain scores over the first 2 postoperative months. At 10 specific time points the "average" pain score following recovery room discharge will be measured using the numeric rating scale. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10= worst imaginable pain. In order to claim that percutaneous cryoneurolysis is superior to usual and customary analgesia, at least one of Outcomes 1 and 2 must be superior while the other at least noninferior.

SECONDARY OUTCOMES:
Opioid consumption | Collected on postoperative days 1, 2, 3, 4, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  Cumulative opioid dose of the previous 24 hours measured in oral oxycodone equivalents
Average Pain | Collected on postoperative days 1, 2, 3, 4, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The "average" pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Worst/maximum Pain | Collected on postoperative days 1, 2, 3, 4, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The "worst" or "maximum" pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Least/lowest/minimal Pain | Collected on postoperative days 3, 7, 14, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The "least" or "lowest" or "minimal" pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Current Pain | Collected on postoperative days 3, 7, 14, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The current pain level at the time of the data collection measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Brief pain Inventory, short form (interference subscale) | Collected on postoperative days 3, 7, 14, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale;(2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale.
First 2 months Brief pain Inventory, short form (interference subscale) | Collected on postoperative days 3, 7, 14, 30, 45 and 60
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale; (2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale. The secondary outcome of greatest interest will be the area under the curve for the interference domain collected over the first two months
Pain with arm raise | Collected on postoperative days 1, 2, 3, 4, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The current pain level at the time of the data collection when the arm is raised measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Awakenings due to pain | Collected on postoperative days 1, 2, 3, 4, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The number of times the patient awoke the previous night due to pain
Post-Traumatic Stress Disorder checklist (PCL-5) | Postoperative day 0 (baseline)
  A 20-item self-report measure reflecting symptoms of post-traumatic disorder validated in military, veteran and civilian populations.
Masking assessment | Postoperative day 7
  Whether or not the patient thinks they received the active cryoneurolysis recorded as "no", "yes", or "unsure"
Phantom Breast Pain (WORST/maximum) | Collected on postoperative days 30 and 45; as well as months 2, 3, 6, 9, and 12
  The "worst" or "maximum" phantom pain level within the operative breast(s) measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain. Phantom pain is defined as pain experienced in breast tissue that is no longer present.
Phantom Breast Pain OCCURRENCES | Collected on postoperative days 30 and 45; as well as months 2, 3, 6, 9, and 12
  The number of times within the previous 24 hours that the participant experienced phantom breast pain. Phantom breast pain is defined as pain experienced in breast tissue that is no longer present.
Phantom Breast Pain DURATION | Collected on postoperative days 30 and 45; as well as months 2, 3, 6, 9, and 12
  The longest duration of phantom breast pain the participant experienced within the previous 24 hours recorded as "seconds", "minutes", or "hours". Phantom breast pain is defined as pain experienced in breast tissue that is no longer present.
Cancer recurrence | First 5 postoperative years queried on postoperative days 30 and 45; as well as months 2, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, and 60
  Any recurrence of the breast cancer in any part of the body
Additional breast surgery | First 5 postoperative years queried on postoperative days 30 and 45; as well as months 2, 3, 6, 9, 12, 24, 36, 48 and 60
  Any additional surgery of the operative breast(s)
Cancer-related therapies | First 5 postoperative years queried on postoperative days 30 and 45; as well as months 2, 3, 6, 9, 12, 24, 36, 48 and 60
  Any additional therapy related to the original mastectomy such as chemotherapy or radiation
Depression screening with the Patient Health Questionnaire (PHQ-2) | Collected on postoperative months 3, 6, 9 and 12
  The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past 2 weeks, scoring each as 0 ("not at all") to 3 ("nearly every day"). The total score therefore ranges from 0-6 with a score of 3 most often used as a cut point when using the PHQ-2 to screen for major depression.
Nociceptive vs neuropathic pain estimation | Collected on postoperative months 6, 9 and 12
  To differentiate nociceptive from neuropathic pain in patients who have a "worst" NRS>0 between 6-12 months, we will administer the self-report Leeds Assessment of Neuropathic Symptoms and Signs pain scale(S-LANSS). A score of 12 or more suggests pain of predominantly neuropathic origin.
Hospitalization duration | Postoperative Days 0-7
  Time from the day of surgery until the day of discharge measured in 1-day increments

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Cedars-Sinai, Los Angeles, California
  - University of California San Diego, San Diego, California
  - University of Florida, Gainesville, Florida
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided